CLINICAL TRIAL: NCT07007208
Title: Biomarkers of the Locus Coeruleus Nucleus: Links With Early Tau Pathology, Cognition and Alzheimer's Disease Risk.
Acronym: Locus-Tau
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/23/0371; 2023-507668-38-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-12; First posted 2025-06-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease
Keywords: PET; MRI; occulometry; locus coeruleus; Alzheimer disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Intervention Model Description: single group with ApoE4 carriers (n=50) and non-ApoE4 carriers (n=50)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- experimental arm (Experimental): TEP exam, MRI exam, oculometry assessment and cognitive tasks
  Interventions: Drug: a positon emission tomography (PET) exam; Other: MRI Contrast; Other: oculometry assessment; Other: cognitive exams

INTERVENTIONS:
Drug: a positon emission tomography (PET) exam — TEP exam using tau-specific tracer ( Flortaucipir, unique dose 360 MBq)
Other: MRI Contrast — Data acquisition will include different sequences (anatomical MRI, resting fMRI). The MRI sequences performed will be anatomical imaging (i.e. T1 imaging, FLAIR), a diffusion sequence, a neuromelanin-sensitive sequence and functional imaging at rest (i.e. "the resting state", which allows the functional connectivity within the so-called "default" network to be assessed).
Other: oculometry assessment — Pupillometry and oculometry will be conducted using an EyeBrain medical device (class IIa). Several cognitive tasks will be submitted to the participant, during which the same measurements will be taken. Different stimuli will be presented on the computer screen (visual scenes, text, geometric shapes) during the eye tracking measurement, and an instruction (cognitive task, such as semantic categorization, free exploration of the gaze, reading, saccade execution) will be associated with each type of stimulus. The successive stimuli will be spaced more than 7 secondes apart in order to allow the pupillary response to the first stimulus to be recorded and then to return to the basal diameter before presentation of the next stimulus.
Other: cognitive exams — Cognitive measures will be acquired during an evaluation session through 6 interactive cognitive exercises. These exercises are developed using tools offered by Covirtua Healthcare.

SUMMARY:
Alzheimer's disease (AD) is characterized by a long-lasting silent phase. Among initial events, emergence of tau pathology in locus coeruleus (LC) brainstem nucleus, well before the one observed in medial temporal cortex, is highly relevant. LC integrity and function can be assessed in vivo with MRI and pupil measures. The current research proposes to evaluate these LC markers in an aged healthy cohort (n=100, with half APOE4 positive) and to relate these markers with cerebral tau pathology, AD risk and cognitive function.

DETAILED DESCRIPTION:
Early tau pathology in the LC may induce dysfunction of the LC-NA system, contribute to initial cognitive decline and possibly be predictive of future AD occurrence. The present project has the following objectives: 1) to relate different biomarkers of LC function measured in vivo with AD risk and future AD occurrence, in order to evaluate their relevance for earliest AD diagnosis, 2) to investigate how LC biomarkers can account for underlying brain tau pathology in asymptomatic older individuals; a related objective will be to validate LC biomarkers as reliable proxies of tau pathology occurrence, and 3) to study the link between LC biomarkers and cognitive performance.

To complete these objectives, the project will evaluate, in healthy older volunteers from the INSPIRE-T cohort (n=100, > 60 years old), biomarkers of LC neuronal integrity, LC-forebrain connectivity, and LC tonic and phasic activity. Additionally, a positon emission tomography (PET) exam will be conducted using tau-specific tracer. Detailed cognitive assessment will also be performed, including assessment of a priori NA-dependent and NA-independent cognitive functions. In the studied cohort (n = 100), half volunteers will be recruited based on genetic AD risk (APOE4 positive) and the other half based on the absence of risk (APOE4 negative).

ELIGIBILITY:
Inclusion Criteria:

* Participant in the INSPIRE-T cohort
* Normal cognitive assessment
* MMSE score ≥ 27 out of 30 (Mini-Mental State Examination)
* Normal visual abilities (in corrected or uncorrected vision)
* Normal motor skills

Exclusion Criteria:

* Subjects with a contraindication to MRI exam
* Subjects with a known allergic reaction to the PET radiopharmaceutical ([18F] Flortaucipir) or any of its excipients
* Subjects with an ophthalmological pathology making oculometric measurements difficult
* Subjects with neurological or psychiatric pathologies

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
diagnostic capabilities of Locus Coeruleus biomarkers for a positive PET-Tau exam | 24 monnths
  The diagnostic capabilities (sensitivity, specificity and AUC) of each of the elements of oculometry (pupillary response, number, latency and amplitude of ocular saccades), functional MRI (LC-hippocampus and LC-prefrontal cortex) and structural MRI (LC intensity) for a positive PET-Tau examination

SECONDARY OUTCOMES:
diagnostic capabilities of Locus Coeruleus biomarkers for a positive PET-Tau exam for the APOe4- groups | 24 months
  The diagnostic capabilities (sensitivity, specificity and AUC) of each of the elements of oculometry (pupillary response, number, latency and amplitude of ocular saccades), functional MRI (LC-hippocampus and LC-prefrontal cortex) and structural MRI (LC intensity) for a positive PET-Tau examination in APOe4- patients
diagnostic capabilities of Locus Coeruleus biomarkers for a positive PET-Tau exam for the APOe4+ groups | 24 months
  The diagnostic capabilities (sensitivity, specificity and AUC) of each of the elements of oculometry (pupillary response, number, latency and amplitude of ocular saccades), functional MRI (LC-hippocampus and LC-prefrontal cortex) and structural MRI (LC intensity) for a positive PET-Tau examination in APOe4+ patients
The relationship between different LC biomarkers | 24 months
  this will be evaluated by correlation and regression. The correlations will be performed both together and separately in the APOe4 status. The impact will be assessed by linear and logistic regression and will also take into account age, gender, and education level.
The link between PET Tau uptake in pupillometry | 24 months
  this will be assessed by the correlation between variations expressed in absolute value or as a proportion of the baseline value and Tau marking, and by regression at 12 and 24 months.. The correlations will be performed both together and separately in the APOe4 status, and the regression will also take into account age, gender, and education level.
The link between PET Tau uptake in oculometry | 24 months
  this will be assessed by the correlation between variations expressed in absolute value or as a proportion of the baseline value and Tau marking, and by regression. The correlations will be performed both together and separately in the APOe4 status, and the regression will also take into account age, gender, and education level.
The link between PET Tau uptake in the structural (neuromelanin) and functional integrity of the LC by MRI | 24 months
  this will be assessed by correlating variations expressed as absolute values or as a proportion of the baseline value with PET Tau, and by regression at 12 and 24 months.
The link between variations in pupillometry | 24 months
  this will be assessed by the correlation between variations expressed in absolute value or as a proportion of the baseline value, and by regression at 12 and 24 months.. The correlations will be performed both together and separately in the APOe4 carrier and non-carrier groups, and the regression will also take into account age, gender, and education level.
The link between variations in occulometry | 24 months
  this will be assessed by the correlation between variations expressed in absolute value or as a proportion of the baseline value, and by regression at 12 and 24 months. The correlations will be performed both together and separately in the APOe4 carrier and non-carrier groups, and the regression will also take into account age, gender, and education level, at 12 and 24 months
The link between variations in the structural (neuromelanin) and functional integrity of the LC by MRI | 24 months
  this will be evaluated by correlation between variations expressed as absolute values or as a proportion of the baseline value and by regression at 12 and 24 months
The relationship between the various LC biomarkers (PET, MRI, pupillometry) and participants' cognitive performance | 24 months
  this will be assessed both at inclusion and at 12 and 24 months, using regressions that take into account age, gender, level of education and APOe4 status.
comparison between APOe4+ and APOe4-: Structural (neuromelanin) and functional integrity of the LC by MRI | 24 months
  this Will be assessed both at inclusion, at 12 months, and at 24 months, through regressions that will take into account age, gender, and education level.
comparison between APOe4+ and APOe4: Cognitive performance | 24 months
  this Will be assessed both at inclusion, at 12 months, and at 24 months, through regressions that will take into account age, gender, and education level.
comparison between APOe4+ and APOe4-: Pupillometry and oculometry | 24 months
  this Will be assessed both at inclusion, at 12 months, and at 24 months, through regressions that will take into account age, gender, and education level.
The reliability of the amplitude of the phasic pupil response during completion of cognitive tasks | 24 months
  This will be validated by intraclass correlation between baseline value and value at one month (test-retest) in a subgroup of 30 participants.
The reliability of the latency of saccadic eye movements during completion of cognitive tasks | 24 months
  This will be validated by intraclass correlation between baseline value and value at one month (test-retest) in a subgroup of 30 participants.
The reliability of the amplitude of saccadic eye movements during completion of cognitive tasks | 24 months
  This will be validated by intraclass correlation between baseline value and value at one month (test-retest) in a subgroup of 30 participants.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No